CLINICAL TRIAL: NCT03216512
Title: A Randomized, Sham-Controlled, Crossover Study to Evaluate the Effects of Noise Cancelling Headphones on Neurocognitive and Academic Outcomes in Children and Adolescents Diagnosed With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Effects of Noise Cancelling Headphones on Neurocognitive and Academic Outcomes in ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bose Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Pro00084739
Record Dates: First submitted 2017-07-06; First posted 2017-07-13 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Proof-of-concept, randomized, within-subject cross-over design.
Who Masked: Participant
Masking Description: The participant won't know whether they are receiving the noise cancelling headphones or the sham control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Noise cancelling headphone first, then sham control headphone (Experimental): This group will use the noise cancelling headphone during the first experimental session as they complete study assessments. They will then return within a week, for experimental session day 2, to complete the same assessments this time using a sham control headphone.
  Interventions: Other: Use of Noise Cancelling Headphones
- Sham control headphone first, then noise cancelling headphone (Experimental): This group will use the sham control headphone during the first experimental session as they complete study assessments. They will then return within a week for experimental session day 2, to redo the same assessments this time using a noise cancelling headphone.
  Interventions: Other: Use of Noise Cancelling Headphones

INTERVENTIONS:
Other: Use of Noise Cancelling Headphones — During the 2 experimental sessions, participants will complete study assessments using either a noise cancelling headphone first (session 1) and then sham control second ( session 2), or vice versa, in the presence of noise distractions.

SUMMARY:
The purpose of this study is to evaluate performance on the Attention Deficit Hyperactivity Disorder ( ADHD) Battery of the Cambridge Automated Neuropsychological Test Battery (CANTAB), including spatial working memory, inhibitory control, and attention while using either a noise cancelling headphone or sham headphone control in the presence of standardized auditory distractors in children and adolescents with ADHD.

DETAILED DESCRIPTION:
This will be a proof-of-concept, randomized, within-subject cross-over design with the administration of noise cancelling headphones or sham headphones on two separate study days. Following screening and a baseline assessment session with no headphones, participants will be assigned to complete each experimental session. During each session, they will undergo the CANTAB and Academic tasks. The order of sessions will be randomized and balanced across participants to be either noise-cancelling headphones first followed by sham headphones; or sham headphones first followed by noise-cancelling headphones. Eligible participants currently taking stimulant medications for ADHD will be asked to stop taking their medication on the day of the baseline visit and during the 2 experimental sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 17 at the time of parental informed consent.
* Male or female.
* Confirmed ADHD diagnosis at screening visit established via MINI-KID (version 7.0.2) administered by a trained clinician.
* Screening ADHD-RS-IV score ≥24.
* Estimated IQ (measured with the KBIT-2) ≥80.
* If currently medicated with a stimulant medication (amphetamine or methylphenidate formulation), off drug on day of Baseline and Experimental Sessions. May resume medication after all assessments are completed on these days.
* Able to follow written and verbal instructions (English) as assessed by the PI and/or study coordinator.
* Able to comply with all testing and requirements.

Exclusion Criteria:

* Current controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis, based on MINI-KID and subsequent clinical interviewing, with significant symptoms including but not limited to post-traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive-compulsive disorder, severe depressive or anxiety disorder, conduct disorder, or other symptomatic manifestations that in the opinion of the Investigator may confound study data/assessments (Participants with clinical history of learning disorders will be allowed to participate as long as the disorder does not impact their ability to participate based on PI judgement).
* Current treatment with any non-stimulant medication for ADHD (e.g., atomoxetine, clonidine, guanfacine).
* Current treatment with other psychoactive drugs.
* Participant is currently considered at risk for attempting suicide by the Investigator, or is currently demonstrating active suicidal ideation or self-injurious behavior, as measured by MINI-KID Suicidality Module C.
* Documented hearing loss.
* Recent history or suspicion (within the past 6 months) of substance abuse or dependence.
* Any other medical condition that, in the opinion of the Investigator, may confound study data/assessments.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants were consented to the study, but failed to meet all inclusion/exclusion criteria
Period: Overall Study
Arm/Group | Noise Cancelling Headphone First, Then Sham Control Headphone | Sham Control Headphone First, Then Noise Cancelling Headphone
Started | 17 | 14
Completed | 17 | 13
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Noise Cancelling Headphone First, Then Sham Control Headphone | Sham Control Headphone First, Then Noise Cancelling Headphone | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.73 (2.30) | 9.52 (2.02) | 9.63 (2.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 11 | 26
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in CANTAB ADHD Battery - Motor Control Task
Description: Compare change from Baseline scores on the Cambridge Automated Neuropsychological Test Battery (CANTAB) ADHD battery with noise cancelling headphones and sham-controls. Results are reported as change from Baseline for each of 4 components of the ADHD battery.
  Motor Control Task: no minimum and maximum values as values are reaction times; positive scores indicate slower reaction times compared to baseline; lower scores indicate faster reaction times compared to Baseline
Time Frame: Baseline, experimental session 1 (3-7 days after baseline), experimental session 2 (3-7 days after experimental session 1)
Measure: Mean (Standard Deviation); unit: reaction time (ms)
Groups:
- Change From Baseline for NC Condition: This is the mean change from Baseline for the NC condition across both arms (NC-Sham and Sham-NC)
- Change From Baseline for Sham Condition: This is the mean change from Baseline for the NC condition across both arms (NC-Sham; Sham-NC)
Arm/Group | Change From Baseline for NC Condition | Change From Baseline for Sham Condition
Number analyzed (Participants) | 31 | 31
reaction time (ms) | -0.033 (0.183) | -0.067 (0.254)

2. Secondary Outcome: Change in Academic Productivity Measures -Math
Description: Compare change from Baseline scores on academic productivity measures (math) - Math Fluency and Calculation Tests (MFACTS) Calculation age standard score; This scale measures an individual's ability to complete age/grade referenced math problems in a set amount of time; higher scores indicate better performance compared to Baseline; standard scores are norm-referenced and have a mean of 100 and a standard deviation of 15. Scores reported here are changes for an individual and can theoretically range from -50 to +50. A higher score indicates better performance in that condition compared to Baseline - ie., better mathematical calculation ability
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Change From Baseline for NC Condition | Change From Baseline for Sham Condition
Number analyzed (Participants) | 31 | 31
score on a scale | 3.77 (8.5) | 0.87 (7.02)

3. Secondary Outcome: Subjective Reports of Experience
Description: Compare the self-reports of noise cancelling headphones versus sham controls - How much did the headphones help you concentrate; self-reported ratings scale with 1 being "not at all" and 10 being "extremely"; higher scores indicate that participants reported better concentration during the session for each condition
Time Frame: Experimental session 1 (3-7 days after baseline), experimental session 2 (3-7 days after experimental session 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- NC Condition; Sham Condition: This is the mean of the self-reported rating for the sessions
Arm/Group | NC Condition | Sham Condition
Number analyzed (Participants) | 31 | 31
score on a scale | 6.53 (2.98) | 6.93 (2.86)

4. Secondary Outcome: Change in Academic Productivity Measures -Reading Comprehension
Description: Compares change from Baseline in Test of Silent Reading and Comprehension (TOSREC) Index score across groups; higher scores indicate better performance compared to Baseline; This scale measures an individual's ability to answer questions about an age/grade referenced reading passage in a set amount of time; higher scores indicate better performance compared to Baseline; Index scores are norm-referenced and can be interpreted similar to standard scores with a mean of 100 and a standard deviation of 15. Scores reported here are changes for an individual and can theoretically range from -50 to +50. A higher score indicates better performance in that condition compared to Baseline - ie., better reading comprehension ability
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Index or Standard Score
Arm/Group | Change From Baseline for NC Condition | Change From Baseline for Sham Condition
Number analyzed (Participants) | 31 | 31
Index or Standard Score | 0.33 (9.68) | -2.27 (9.74)

5. Primary Outcome: Change in CANTAB ADHD Battery - Spatial Working Memory Task
Description: Compare change from Baseline scores on the Cambridge Automated Neuropsychological Test Battery (CANTAB) ADHD battery with noise cancelling headphones and sham-controls. Results are reported as change from Baseline for each of 4 components of the ADHD battery.
  Spatial Working Memory Task: no minimum and maximum values as values are number of errors; higher (positive) scores indicate more errors compared to Baseline
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Change From Baseline for NC Condition | Change From Baseline for Sham Condition
Number analyzed (Participants) | 31 | 31
errors | -3.28 (7.66) | -3.48 (9.26)

6. Primary Outcome: Change in CANTAB ADHD Battery - Stop Signal Reaction Time Task
Description: Compare change from Baseline scores on the Cambridge Automated Neuropsychological Test Battery (CANTAB) ADHD battery with noise cancelling headphones and sham-controls. Results are reported as change from Baseline for each of 4 components of the ADHD battery.
  Stop Signal Reaction Time Task: no minimum and maximum values as values are reaction times; higher scores indicate worse performance compared to Baseline
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: reaction time (ms)
Arm/Group | Change From Baseline for NC Condition | Change From Baseline for Sham Condition
Number analyzed (Participants) | 31 | 31
reaction time (ms) | 117.56 (95.28) | 78.41 (26.99)

7. Primary Outcome: Change in CANTAB ADHD Battery - Rapid Visual Processing Task
Description: Compare change from Baseline scores on the Cambridge Automated Neuropsychological Test Battery (CANTAB) ADHD battery with noise cancelling headphones and sham-controls. Results are reported as change from Baseline for each of 4 components of the ADHD battery.
  Rapid Visual Processing Task: no minimum and maximum values as values are number of correct hits; higher scores indicate better performance compared to Baseline
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: correct hits
Arm/Group | Change From Baseline for NC Condition | Change From Baseline for Sham Condition
Number analyzed (Participants) | 31 | 31
correct hits | -0.013 (0.079) | 0.001 (0.081)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of Screening/Enrollment until the last experimental session, which constituted the end of the study, which was on average 4 weeks from the time of Screening
Groups:
- Noise Cancelling Headphones: This arm is during sessions when participants received noise cancelling headphones
- Sham Control Headphones: This arm is during sessions when participants received sham control headphones
Arm/Group | Noise Cancelling Headphones | Sham Control Headphones
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03216512/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT03216512/Prot_SAP_001.pdf